CLINICAL TRIAL: NCT05038865
Title: Oral Health Related Quality of Life - The Effect of Malocclusions, Gender, Socioeconomic Differences and Orthodontic Treatment Among Adolescents
Brief Title: The Effect of Malocclusions on Oral Health Related Quality of Life
Status: Recruiting | Type: Observational
Sponsor: Malmö University (Other)
Collaborators: Region Östergötland (Other); Folktandvården Stockholms län AB (Other Government)
Responsible Party: Principal Investigator, Mikael Sonesson, Dr, Malmö University
Other Study IDs: 2020-05319
Record Dates: First submitted 2021-02-22; First posted 2021-09-09 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Malocclusion; Quality of Life; Orthodontics; Adolescent; Socioeconomic Factors
MeSH Terms: conditions — Malocclusion | interventions — Orthodontics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Malocclusion group: 500 12-19 year olds with malocclusion, defined as IOTN-DHC grade 3, 4 or 5. The adolescents are consecutively recruited new patients at three orthodontic centers; Center for Orthodontics and Pediatric Dentistry, Norrköping, Public Dental Service Östergötland; Department of Orthodontics, Folktandvården Stockholms län AB, Folktandvården Eastmaninstitutet, Stockholm, Sweden and Department of Orthodontics, Malmö University, Malmö, Sweden. Patients are examined at the first visit at the orthodontic department, before any orthodontic treatment is begun.
  Interventions: Other: Malocclusion and Orthodontic Treatment
- No malocclusion group: 175 12-19 year olds without malocclusion, defined as IOTN-DHC grade 1 or 2. Patients are consectively recruited adolescents examined at their general dentistry clinic.

INTERVENTIONS:
Other: Malocclusion and Orthodontic Treatment — Group 1 is exposed to malocclusion and orthodontic treatment. However, the inclusion in the study does not affect the treatment since it is an observational study.
  The exposure of group 2 is no malocclusion, no orthodontic treatment.
  Groups: Malocclusion group

SUMMARY:
Malocclusions in adolescents may affect oral health related quality of life. The study aims at;

1. Evaluating two instruments measuring oral health related quality of life; "Child Perceptions Questionnaire 11-14" (CPQ 11-14) short form and "Psychosocial Impact of Dental Aesthetics Questionnaire" (PIDAQ).
2. Comparing differences in oral health related quality of life in;

   1. adolescents with different types of malocclusion and without malocclusions
   2. individuals of different genders and socioeconomic status
3. Longitudinally evaluating differences in oral health related quality of life;

   1. before, during and after orthodontic treatment
   2. in untreated individuals (without malocclusion) over time

DETAILED DESCRIPTION:
The individuals that are to be recruited to the study are;

Malocclusion group; 500 12-19 year olds with malocclusion, examined at their specialist orthodontic clinic.

No malocclusion group; 175 12-19 year olds without malocclusion, examined at their general dentistry clinic.

All patients will also answers two questionnaires (in Swedish) measuring oral health related quality of life; CPQ 11-14 short form (Jokovic 2006, Dimberg 2019) and PIDAQ (Klages 2006, Göranson 2020). Randomization will ensure that half of the study participants will begin with CPQ 11-14 short form and then PIDAQ, while half of the participants will answer the questionnaires in the reverse order. The questionnaires will be answered in a calm environment in the dental clinic.

All patients will have five standardized intraoral photographs taken. These photographs are already routinely taken at the specialist orthodontic clinics, but is taken in addition to routine procedure at the general dentistry clinic. To determine presence of malocclusion and orthodontic treatment need, two orthodontic indices will be used; ICON (Daniels 2000) and IOTN (Brook 1989). Assessments will be based on intraoral photographs, clinical measurements and pre-existing dental x-rays.

Also, patients will be grouped based on their type of malocclusion using the following diagnoses;

* Enlarged overjet (≥ 6 mm) with or without incomplete lip closure
* Anterior cross bite (One or more incisors)
* Deep bite (≥ 2/3 lower incisor coverage)
* Frontal open bite (≤0 mm)
* Lateral cross bite (two or more teeth, with our without lateral guidance)
* Upper or lower arch anterior spacing (largest gap between two neighbouring teeth between canine and canine ≥ 2 mm)
* Upper or lower arch anterior crowding (≥ 3 mm lack of space canine to canine)

As the study is of longitudinal design, the questionnaires will be answered and the photographs will be taken on several occasions. For the malocclusion group, the time points will be as following;

* T0- at the initial examination at the specialist orthodontic clinic, before orthodontic treatment is begun
* T2- One year into the orthodontic treatment
* T3- Two months after the orthodontic treatment has been completed
* T4- One year after the orthodontic treatment has been completed.

The no malocclusion group will be examined the same number of times and at the same time intervals as the malocclusion group.

Information about DMFT/S (decayed, missing, filled, teeth/surfaces will be gathered from the dental records. Orthodontic extractions will be noted. To be able to determine socioeconomic differences, information about socioeconomic status of the individual study participants will be gathered from the Statistics Sweden.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents 12-19 years of age with malocclusion (IOTN grade 4 and 5) referred to specialist orthodontic clinics
* Adolescents 12-19 years of age without malocclusion (IOTN grad 1, 2 or 3) at general dentistry clinics

Exclusion Criteria:

* Previous orthodontic treatment
* Cleft lip and palate
* ASA ≥ III
* Intellectual and/or physical inability to answer questionnaires

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Malocclusion group 500 12-19 year olds with malocclusion, defined as IOTN-DHC grade 3, 4 or 5. The adolescents are consecutively recruited new patients at three orthodontic centers; Center for Orthodontics and Pediatric Dentistry, Norrköping, Public Dental Service Östergötland; Department of Orthodontics, Folktandvården Stockholms län AB, Folktandvården Eastmaninstitutet, Stockholm, Sweden and Department of Orthodontics, Malmö University, Malmö, Sweden. Patients are examined at the initial examination at the orthodontic department, before any orthodontic treatment is begun.
  No malocclusion group 175 12-19 year olds without malocclusion, defined as IOTN-DHC grade 1 or 2. Patients are consectively recruited adolescents examined at their general dentistry clinic.
Sampling Method: Probability Sample
Enrollment: 675 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Oral Health Related Quality of Life measured with Child Perceptions Questionnaire 11-14 short form- change before and after orthodontic treatment and at matched time points in an untreated population | At start of study, 1 year after start of study, at study completion (an average of 2.5 years), 1 year after study completion
  Child Perceptions Questionnaire (CPQ) 11-14 short form is a common instrument measuring Oral Health Related Quality of life (OHRQoL) in children and adolescents. It is a generic instrument, measuring all aspects of OHRQoL.
Oral Health Related Quality of Life measured with Psychosocial Impact of Dental Aesthetics Questionnaire - change before and after orthodontic treatment and at matched time points in an untreated population | At start of study, 1 year after start of study, at study completion (an average of 2.5 years), 1 year after study completion
  Psychosocial Impact of Dental Aesthetics (PIDAQ) is an instrument measuring orthodontic specific aspects of OHRQoL.

CONTACTS AND LOCATIONS:
Overall Officials: Mikael Sonesson, PhD, Principal Investigator — Malmö University
Locations (3):
- Sweden (3):
  - Mikael Sonesson, Malmo, Skåne County
  - Folktandvården Östergötland, Linköping
  - Eastman Institutet Ortodonti, Stockholm

REFERENCES:
- [Background] Jokovic A, Locker D, Guyatt G. Short forms of the Child Perceptions Questionnaire for 11-14-year-old children (CPQ11-14): development and initial evaluation. Health Qual Life Outcomes. 2006 Jan 19;4:4. doi: 10.1186/1477-7525-4-4. PMID 16423298
- [Background] Dimberg L, Lennartsson B, Bondemark L, Arnrup K. Validity and reliability of the Swedish versions of the short-form Child Perceptions Questionnaire 11-14 and Parental Perceptions Questionnaire. Acta Odontol Scand. 2019 Nov;77(8):630-635. doi: 10.1080/00016357.2019.1634282. Epub 2019 Jul 3. PMID 31267808
- [Background] Klages U, Claus N, Wehrbein H, Zentner A. Development of a questionnaire for assessment of the psychosocial impact of dental aesthetics in young adults. Eur J Orthod. 2006 Apr;28(2):103-11. doi: 10.1093/ejo/cji083. Epub 2005 Oct 28. PMID 16257989
- [Background] Goranson E, Norevall LI, Bagesund M, Dimberg L. Translation and validation of the Swedish version of the Psychosocial Impact of Dental Aesthetics Questionnaire (PIDAQ) for adolescents. Acta Odontol Scand. 2021 May;79(4):241-247. doi: 10.1080/00016357.2020.1823014. Epub 2020 Oct 7. PMID 33026890
- [Background] Daniels C, Richmond S. The development of the index of complexity, outcome and need (ICON). J Orthod. 2000 Jun;27(2):149-62. doi: 10.1093/ortho/27.2.149. PMID 10867071
- [Background] Brook PH, Shaw WC. The development of an index of orthodontic treatment priority. Eur J Orthod. 1989 Aug;11(3):309-20. doi: 10.1093/oxfordjournals.ejo.a035999. PMID 2792220
- [Derived] Goranson E, Sonesson M, Gullbrand M, Isberg PE, Dimberg L. The Reliability and Validity of Intraoral Photographs in Assessing Orthodontic Treatment Need. Orthod Craniofac Res. 2025 Jun;28(3):474-484. doi: 10.1111/ocr.12896. Epub 2025 Jan 13. PMID 39803929